CLINICAL TRIAL: NCT06681233
Title: A Feasibility Study of a Novel Cone-Beam CT Approach for Image Guided Radiotherapy in Cancer Patients
Brief Title: Feasibility Study of CBCT for IGRT in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2023-04
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancers; Breast Cancer; Thoracic Cancers; Liver Cancer; Genito Urinary Cancer; Gastrointestinal Cancers
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Liver Neoplasms; Urogenital Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-site feasibility study designed to generate data evaluating the quality and applicability of the HyperSight on-couch high-performance CBCT imaging technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HyperSight Imaging Arm (Experimental)
  Interventions: Device: Comparison of HyperSight CBCT imaging to conventional CBCT imaging.

INTERVENTIONS:
Device: Comparison of HyperSight CBCT imaging to conventional CBCT imaging. — Participants will receive their daily radiation treatment on a radiation therapy system equipped with HyperSight CBCT imaging. For at least 1 and up to 3 treatment fractions, participants will receive their daily radiation treatment on a system equipped with conventional CBCT imaging.

SUMMARY:
Cone beam computed tomography (CBCT) is an imaging technology that is incorporated into many modern radiation therapy systems. The quality of conventional CBCT is good enough to align patients for their daily radiation therapy but CBCT images have poor contrast and are susceptible to imaging artefacts that limit their usability for other tasks in the radiation therapy workflow.

Varian Medical Systems, the sponsor of this study, has developed new CBCT imaging technology called HyperSight that so far has demonstrated increased image quality compared with conventional CBCT images. This new HyperSight CBCT imager has previously been built into Varian Halcyon and Ethos treatment machines, where the imager is enclosed in a ring that rotates around the patient. Now, HyperSight has been built into a Varian treatment machine, called TrueBeam, where the imager is mounted on a C-shaped arm that rotates around you to acquire an image.

This study is being done to evaluate the image quality of HyperSight CBCT compared to conventional CBCT images, and to determine whether HyperSight CBCT can improve the process of delivering radiation treatments.

The goal of this study is to collect images from this new HyperSight-TrueBeam CBCT imager from a variety of patients and locations in the body. The images will be analyzed to determine whether their quality is high enough to use for tasks other than positioning patients for treatment. For example, the study will determine whether the HyperSight images could be used to calculate a radiation plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18
2. Patient is receiving radiation therapy for head and neck, thorax, liver, breast, genitourinary, or gastrointestinal malignancies
3. A CBCT acquisition for localization is standard of care for the radiation therapy treatment plan being delivered

Exclusion Criteria:

1. Patient has ECOG Performance Status ≥3.
2. Patient is wheelchair bound.
3. Patient has a life expectancy <3 months.
4. Patient is unwilling or unable to provide informed consent to participate in the study.
5. Patient is pregnant or has plans for pregnancy during the period of treatment.
6. Patient is part of a vulnerable population (per ISO 14155:2020, "individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response"). This includes prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of Image Contrast Resolution | End of radiation treatment at 9 weeks.
  The difference in contrast resolution will be evaluated between a standard CBCT image, a CBCT image acquired using HyperSight technology, and a standard fan-beam CT acquired as part of the treatment simulation and planning process
Comparison of Image Uniformity | End of radiation treatment at 9 weeks.
  The difference in image uniformity will be evaluated between a standard CBCT image, a CBCT image acquired using HyperSight technology, and a standard fan-beam CT acquired as part of the treatment simulation and planning process.
Qualitative Image Comparison | End of radiation treatment at 9 weeks.
  Qualitative comparison of HyperSight CBCT to conventional CBCT to determine preferred imaging for patient localization for daily treatment. Clinician observers will rank their preference using a 5-point Likert scale, where 1 represents strong preference of one imaging modality and 5 represents strong preference for the other modality.

SECONDARY OUTCOMES:
Reduction of Metal Artifacts | End of radiation treatment at 9 weeks.
  In patients with a metal implant in the imaging field, the volume [cubic centimeters] of the metal artefact will be compared between a standard CBCT image, a CBCT image acquired using HyperSight technology, and a standard fan-beam CT acquired as part of the treatment simulation and planning process.
Imaging Time for Large Treatment Volumes | End of radiation treatment at 9 weeks.
  For participants where multiple conventional CBCTs must be acquired and stitched together to capture the entire treatment field, the time [seconds] required for the overall imaging session will be recorded and compared between HyperSight CBCT and conventional CBCT.
Imaging Time for Breath Hold Imaging | End of radiation treatment at 9 weeks.
  For participants who undergo breath-hold imaging, the time [seconds] required for the overall imaging session will be recorded and compared between HyperSight CBCT and conventional CBCT.
Patient Tolerance of Breath Hold Imaging | End of radiation treatment at 9 weeks.
  For participants who undergo breath-hold imaging, the total number of individual breath-holds required for a complete image acquisition will be recorded and compared between HyperSight CBCT and conventional CBCT.
Feasibility of HyperSight CBCT for Treatment Planning | End of radiation treatment at 9 weeks.
  For anatomical regions where there are limited anatomical deformations expected between image acquisitions, the radiation doses calculated for individual anatomical structures in a participant's treatment plan, which is based on their fan-beam simulation CT, will be compared to doses for the same structures after re-calculating the dose distribution for the same treatment plan using both the HyperSight CBCT and conventional standard CBCT.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No